CLINICAL TRIAL: NCT03676309
Title: Efficacy and Safety of Nutraceuticals (Bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg) in Patients With Diabetes Mellitus Type II and Dyslipidemia.
Brief Title: Efficacy and Safety of Nutraceuticals in Patients With Diabetes Mellitus Type II and Dyslipidemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Villa dei Gerani (Other)
Collaborators: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Capomolla Antonio, Division Director, Villa dei Gerani
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PON03PE_00078_2
Record Dates: First submitted 2018-09-10; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2; Nutritional and Metabolic Diseases; Vascular System Injury; Therapy-Related Morphologic Change
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Nutritional and Metabolic Diseases; Vascular System Injuries | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: Experimental drawing Phase II prospective, randomized, comparative, vs placebo study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): placebo tablet twice a day twenty minutes before main meals, for 12 weeks,
  Interventions: Drug: Placebo Oral Tablet
- nutraceutical oral capsule (Active Comparator): nutraceutical oral capsule 920 mg twice a day for 12 weeks
  Interventions: Drug: Nutriceutical Oral Capsule,

INTERVENTIONS:
Drug: Nutriceutical Oral Capsule, — nutraceutical 920 mg (Bergamot 450 mg, Gymnema (400 mg, Phaseolamine 30 mg, Olea Europaea 10 mg) twice day , 12 weeks
  Arms: nutraceutical oral capsule
Drug: Placebo Oral Tablet — placebo tablet twice a day twenty minutes before main meals, for 12 weeks,
  Other Names: placebo tablet
  Arms: placebo

SUMMARY:
The presence of dyslipidemia, is a significant cardiovascular risk factor. This factor, however, determines the three-fold increase in cardiometabolic risk when an isolated or mixed dyslipidemia is associated with the presence of diabetes mellitus. Diabetes mellitus is a metabolic alteration resulting in a decrease in insulin secondary to reduced availability of this hormone or an impediment to its normal action or a combination of these factors. . Under normal conditions, the vascular endothelium responds to short-term increases in flow by releasing NO and other endothelium-dependent relaxing factors that dilate the artery. Flow-mediated dilation(FMD) is impaired in atherosclerotic coronary arteries. The supplementation with polyphenols of olive leaves, bergamot extract, gymnema sylvatic extract (gymnemic acid) and phaseolamin (bean protein) significantly improves the glico-lipid balance through an improvement in liver function, an inhibition to more levels of lipid metabolism .

Recently, it has been documented how the polyphenolic fraction extracted from bergamot (BPF) administered orally both in animal models with induced hyperlipidemia diet, and in patients with metabolic syndrome, produces a significant and substantial reduction of serum cholesterol, triglycerides and blood levels of glucose. This effect was accompanied by an important improvement in vascular reactivity in patients with hyperlipidemia and high blood sugar, suggesting the potential protective role of BPF in patients with metabolic syndrome and elevated cardiovascular risk.

Oleuropeina (Olea Europaea) is also characterized by a peculiar polyphenolic profile. Both fruits and leaves, thanks to their cardioprotective activity, are used as antihypertensive agents and in the treatment of vascular disorders. The gymnemic acid (glycosidic triterpene), extracted from the leaves of Gymnema Sylvestre, is the representative element of the plant. Thanks to its presence in the phytocomplex, it carries out a hypoglycaemic action through two main mechanisms: inhibition of intestinal sugar absorption and increased metabolic transformation of glucose at the cellular level.

To better define the interrelations of systemic CRFs, FMD, and effects of chronic nutraceutical supplements we performed clinical evaluations and ultrasound measurements of the flow and diameter responses to forearm cuff occlusion in a large, well characterized community-based cohort.

DETAILED DESCRIPTION:
Primary end point Effectiveness To demonstrate in diabetic patients,the effectiveness of nutraceuticals (bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg) to reduce total and LDL cholesterol.

Secondary end points To demonstrate in diabetic patients,the effectiveness of nutraceuticals (bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg) to improve Endothelial function evaluated with vascular Doppler color echo; CHARACTERISTICS OF THE POPULATION diabetic patients in optimized medical therapy and increased plasma levels of total and LDL cholesterol EXPERIMENTAL DESIGN AND METHODOLOGY OF RESEARCH Experimental drawing Phase II prospective, randomized, comparative, vs placebo study Sample size Literature data show that total cholesterol levels> 200 mg / dl and LDL> 130 mg//dl have an increased cardiovascular risk in subjects with diabetes mellitus; in the Calabrian people the Health Examination Survey conducted in 2012, showed the following average values: total cholesterolemia 233 +/- 45 mg /dl for men and 238 +/- 40 mg / dl for women; while for LDL cholesterol the mean values are respectively 151 +/- 30 mg / dl in humans and 148 +/- 35 mg / dl in women. In these subjects the doubling of the statin dosage contributes to a further reduction of plasma levels by about 6%; the hypothesis not evaluated is that the integration with nutraceuticals (bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg) in patients with optimized therapy, involves reduction of plasma levels> 6% HYPOTHESIS N =2(1600)/(196)*6,2= 3200/196*6.2= 88 The study will be performed with the enrollment of 88 diabetic patients, Eligible patients will be of both sexes, and naïve patients on nutraceutical (920 mg), consequently recruited.

Patients using randomization tab will be randomized 1: 1 to treatment with active substance versus placebo. Investigators may not be aware of the sequence in which the treatments will be assigned nor foresee the next assignment in any way.

TIMING OF THE STUDY The duration of the study will be 12 weeks after recruitment. After signing the informed consent, previously approved by the Ethics Committee, the subjects can fully enter the study. Each patient must make three visits: SEL (selection visit); V01 (initial visit); TERM (final visit). Excluding the patient's inclusion visit (V01), each visit will take place in the morning and each patient will be studied at the same time of day, between 8.00 am and 12.00 am, during the study (± 2 hours).

The treatment is always accompanied by main meals. The first administration in naïve patients on Nutraceuticals will be done under the supervision of the staff involved in the study. Patients will then be reviewed at 4 and 12 weeks after recruitment.

ANALYTICAL PRESENTATION OF THE PROCEDURES TO BE PERFORMED Before signing informed consent, patients will be informed about the rationale of the study, the objective and the procedures of the study itself. All the subjects can refuse to participate, or they can interrupt the participation at any time.

The study will be conducted in accordance with the protocol, Good Clinical Practice (GCP) and according to the regulatory principles of application.

Selection visit During the selection visit (SEL), all patients are subjected to the following evaluation.

* Collection of informed consent by the principal investigator;
* Complete medical documentation on anthropological characteristics and clinical anamnesis (including any chronic treatments, or in the case of women, of contraceptive measures), and assessment of the presence of inclusion and exclusion criteria;
* Data collection: weight, height, Body Mass Index calculation, Systolic Blood Pressure and Diastolic Blood Pressure measurements (mean arterial pressure) using automatic meters, and 12-lead electrocardiogram;
* Blood chemistry tests (total ,LDL and HDL cholesterol, glycemia, triglycerides, creatinine, Glutamic Oxaloacetic Transaminase(GOT), Glutamic Piruvate Transaminase (GPT), , potassium(K), Sodium (Na) uricemia and blood count, hb glycated blood sugar, C-reactive Protein );
* Electrocardiogram
* cardiac Eco-color - doppler (evaluation of the systolic and diastolic function indices)
* Non-invasive study of endothelial function (vascular arterial Doppler )
* Ergometric test
* Six minutes walking test
* Questionnaire on quality of life SF 36
* Pregnancy test in women of childbearing age

All laboratory results and pregnancy tests are checked before enrolling the patient in the study:

If the result of these evaluations:

A) Does not meet the inclusion criteria, the investigator must:

* Document all the interview and the occurrence of adverse events;
* Draw up the examination and a physical exam including weight, height and measurements of systolic and diastolic pressures;
* Examine all the results of blood chemistry and biochemical tests; Document the reasons why the patient is not included in the study. Complete the CRF (case report Forms) of the trial. B) Satisfy the inclusion criteria (and if exclusion criteria do not appear), a blood sample will be collected.

Therefore, the patients eligible for the study will be recruited and treated with:

* nutraceuticals (bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg)
* Placebo Patients will take part in the study by double daily administration, before main meals. The first administration always takes place in the presence of personnel involved in the study VISIT 1 (4 WEEKS) Patients enrolled are promptly informed on the dosage of treatment, on compliance with treatment and on the need to evaluate its effectiveness after four weeks (± 3 days): V01.

During the 4-week visit (V01), patients undergo:

* Collection of any symptoms related to gastrointestinal disorders
* Blood sampling: Blood chemistry tests (total cholesterol, LDL and HDL cholesterol, glycemia, triglycerides, creatinine, GOT , GPT, Na, K, uricemia and blood count, hb glycated blood sugar, insulin, CrP )
* Objective examination
* Detection of vital parameters (blood pressure, heart rate)
* Interview on adverse events, if present, and concomitant changes to the assumption of treatment
* Restitution of the drug and calculation of unused capsules to assess patient compliance
* Reporting in the CRF of the number of unused and returned capsules
* Delivery of the drug. FINAL VISIT (TERM)

During the final visit (TERM), made twelve weeks after enrollment (± 3 days), patients undergo the evaluation of:

* Data collection: weight, height, BMI calculation, SBP and DBP measurements (mean arterial pressure) using automatic meters, and twelve-lead electrocardiogram;
* Blood chemistry tests (total cholesterol, LDL and HDL cholesterol, glycemia, triglycerides, creatinine,GOT, GPT, Na, K, uricemia and blood count, hb glycated blood sugar, insulin,CrP)
* Electrocardiogram
* Cardiac Eco-color doppler (evaluation of the indices of systolic and diastolic function)
* Non-invasive study of endothelial function (vascular arterial Doppler)
* Ergometric test
* Six minutes walking test
* Questionnaire on quality of life SF 36
* Collection of any symptoms related to gastrointestinal disorders
* Interview on adverse events, if present, and concomitant changes to the assumption of treatment
* Restitution of the drug and calculation of unused capsules to assess patient compliance
* Reporting in the CRF of the number of unused and returned capsules. EARLY TERMINATION OF THE STUDY After informing the Ethics Committee and the Health Authorities, the person who took part in the study may decide to stop the study before the deadline.

Two copies of the written consent will be dated and signed by the investigator. All data will be collected in the case report (CRF) INTERRUPTION OF THE TREATMENT Withdrawal and interruption of a patient's study A patient can withdraw from the study at any time.

The treatment may be prematurely and permanently interrupted by the investigator for one or more of the following reasons:

* Patient refusal to continue the study
* Principle of an adverse event, which represents an important risk to the patient according to the investigator or requires the prescription of treatments that are not considered concomitant in the protocol.
* Treatment not tolerated
* Any clinical event that requires treatment interruption.
* Any clinical event that requires a type of treatment that is incompatible with the study.
* Pregnancy Procedures

In case of premature interruption of treatment:

- the investigator must document the reason (s) and the exact time of the interruption of the study in the CRF and in the patient's record. If more than one reason is given, the investigator must indicate the main one.

In the case of a premature withdrawal from the study due to an adverse event (an event requiring immediate notification or not), the investigator must collect all the information related to the event. If necessary, the information is put together later.

- During the final follow-up visit, the investigator must:

* Draw up the interview on the occurrence of an adverse event and on the changes in the treatment and the respective doses;
* Perform objective examination (including weight, height, systolic and diastolic blood pressure);
* Perform a twelve-lead ECG
* Carry out a withdrawal for renal and hepatic function, possibly fasting blood count;
* Recover the remaining capsules and report in the CRF the number of unused and returned capsules;
* Document the date of the first and last administration taken;
* Estimate patient compliance with treatment between the final and previous visits.

ADVERSE EVENTS AND ADVERSE REACTIONS Serious adverse event and adverse drug reactions The European legislation on pharmacovigilance was amended with the adoption in 2010 of EU Regulation 1235/2010, whose application is operational from 2 July 2012, and of Directive 2010/84 / EU, in force since 21 July 2012.

Collection and notification, by the individual Investigators and by the Promoter, of adverse events / adverse reactions occurred to patients enrolled in clinical trials with medicinal products for human use. For the definition of serious and non-serious adverse events, refer to the Standards of Good Clinical Practice of the PATIENT TREATMENTS Treatment management There is only one treatment period, and the formulation of the drug is in capsule form. The treatment is provided directly by the investigator at the end of each scheduled visit. Patients will take the product in a single daily dose after one of the main meals.

Delivery of treatment

Patients will be divided into two groups:

Group 1 composed of 45 enrolled subjects who will receive placebo bis in die, twenty minutes before the main meals; Group 2 composed of 45 subjects enrolled with type II diabetes mellitus and hypercholesterolemia without hypertriglyceridemia who will receive a double administration of nutraceuticals (bergamot 450 mg, Gymnema (400 mg, Phaseolamin 30 mg, Olea Europaea 10 mg) mg with the cadences described for group 1; Previous and concurrent treatments All details on previous and concurrent treatments must be collected by the investigator in an appropriate form in the CRF. It will be the duty of the investigator to always evaluate that concomitant and / or previous treatments are authorized and included in the inclusion criteria.

STATISTICAL ANALYSIS All values are expressed as mean +/- Standard deviation. The values of the selected variables in perspective mode will be expressed as mean +/- standard deviation (parametric variables) or median (non parametric variables). To compare the differences between the study groups, correlation analysis, t-test for samples, independent, chi-square test, frequency tables, cross tables and tables for multiple / dichotomous responses will be used. A probability value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the patient
* Fasting plasma glucose ≥ 126 mg / dl (7 mmol / l);
* Hypercholesterolemia (LDL cholesterol ≥ 130 mg / dl), with or without hypertriglyceridemia (> 175 mg / dl);
* Medical therapy stabilized for 4 months. For women of reproductive age, enrolled in the study, the non-occurrence of pregnancy must be guaranteed.

All concomitant treatments should have started at least 3 months before the start of the study and should be kept at a constant dose throughout the study.

Exclusion Criteria:

* Positive pregnancy test (βGCH), made at the selection visit (SEL) or in any case doubtful, pregnant women, lactating women, women of childbearing age who do not use estrogens or progestogens or intrauterine contraceptive methods;
* Patients with severe gastrointestinal disorders with possible influence of the drug on electrolytes and absorption;
* Patients with severe kidney disease (GFR 30 mL / min / 1.73 m2),
* Patients with liver disease or obstructive disorders of the biliary tract, with or without complications (chronic hepatitis, cirrhosis, etc.), or with GOT or GPT at the upper limits of 3 times the laboratory reference values;
* History of alcoholism or drug abuse;
* Clinical history of serious illness that can in some way interfere with the conduct of the study, infections and neoplasms;
* History of psychiatric disorders, major depression, or suicide attempts;
* Patients with HIV or taking HIV medications
* Presence of low-threshold myocardial ischemia
* Presence of heart failure of class III and IV NYHA (New York Heart Association)
* Patients with current infections
* Valve prosthesis patients;
* Patient with atrial fibrillation;
* Patients with contraindication to physical exercise;

Min Age: 30 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
colesterol | "day 0" , "month 1", "month 3"
  change cholesterol,

SECONDARY OUTCOMES:
Endothelial function | "day 0" , "month 3"
  change shear rate
Endothelial function | "day 0" , "month 3"
  change shear rate after ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Capomolla Antonio, MD, Principal Investigator — Villa dei Gerani
Locations (1):
- Capomolla Antonio, Monterosso Calabro, VV, Italy

IPD SHARING:
Plan to Share IPD: No